CLINICAL TRIAL: NCT05676827
Title: Assessment of the Relationship Between Pain, Central Sensitization and Psychoemotional State in Patients With Chronic Masticatory Muscle Pain
Brief Title: Pain, Central Sensitization and Psychoemotional State in Patients With Chronic Masticatory Muscle Pain
Status: Enrolling by invitation | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Smardz, Investigator, Wroclaw Medical University
Other Study IDs: WMU1/2022
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: TMD; Masticatory Muscle Pain
Keywords: TMD, masticatory muscle pain, central sensitization
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Participants with masticatory muscle pain lasting for over 3 months.
  Interventions: Diagnostic Test: Diagnostic Criteria for Temporomandibular Disorders Clinical Examination; Diagnostic Test: Blood test
- Control group: Participants without masticatory muscle pain in last 6 months.
  Interventions: Diagnostic Test: Diagnostic Criteria for Temporomandibular Disorders Clinical Examination; Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Diagnostic Criteria for Temporomandibular Disorders Clinical Examination — Clinical examination made by experienced dentists (minimum 5 years of practice) and trained and calibrated in accordance with the protocol available on the DC/TMD.
Diagnostic Test: Blood test — Blood samples will be tested to investigate two polymorphisms of genes encoding proteins for serotonin receptors HTR2A - rs4941573 in intron 3 and dopamine DRD3 - rs6280 (Ser9Gly) and levels of serotonin, dopamine, Gamma-aminobutyric acid (GABA), Tumor Necrosis Factor α (TNF-α), CGRP, SERT, interleukin 1B, interleukin 6, interleukin 8, interleukin 10 and interleukin 17A.

SUMMARY:
The aim of this study is to investigate the relationship of psychological aspects, selected blood parameters, pain, central sensitization, and muscle electromyography activity in patients with chronic masticatory muscle pain.

DETAILED DESCRIPTION:
In this prospective cohort study, the study group will consist of 51 people with masticatory muscle pain lasting longer than 3 months, while the control group will involve 51 people without such disorder.

Muscle type of temporomandibular disorders will be diagnosed on the basis of validated and standardized DC/TMD protocol.

Additionally potential headaches will be assessed according to the ICHD-3, since coexistence of chronic masticatory muscle pain and headache is often observed.

Psychological aspects will be analyzed using validated questionnaires regarding depression (PHQ-9), anxiety (GAD-7), perceived stress (PSS-10), satisfaction with life (SWLS), type D personality (DS-14) and coping with stress (Mini-COPE). Central Sensitization will be assessed using the Central Sensitization Inventory. Following blood substances will be assessed: serotonin, dopamine, Gamma-aminobutyric acid (GABA), Tumor Necrosis Factor α (TNF-α), CGRP, SERT, interleukin 1B, interleukin 6, interleukin 8, interleukin 10 and interleukin 17A. Additionally two polymorphisms of genes encoding proteins for serotonin receptors HTR2A - rs4941573 in intron 3 and dopamine DRD3 - rs6280 (Ser9Gly) will be analyzed.

Pain assessment will be done using a validated and standardized questionnaire regarding chronic pain (GCPS) and an algometer and will include the measurement of pressure pain threshold in masseter and temporal muscles. In addition, potential autonomic disorders will be assessed using Autonomic Symptoms Questionnaire proposed by Low. Electromyographic muscle activity will be assessed by tetany test. The results of the study will allow for deeper understanding of the complex nature of orofacial pain of muscle origin and its connection with the mechanism of central sensitization, headache and muscle electromyographic activity. Measurement of blood parameters will provide more accurate information on the pathophysiology of these disorders and the use of validated questionnaires will provide valuable information about the mental state of patients.

ELIGIBILITY:
Inclusion Criteria for study group:

* Masticatory muscle pain for at least 3 months, based on DC/TMD, at least 18 y.o

Exclusion Criteria:

* severe neurological or psychiatric diseases, use of drugs that may affect the neuromuscular system, alcohol or drug addiction, cancer or pregnancy, previous head surgery

Inclusion criteria for control group:

* no pain in masticatory muscles, age of at least 18 y.o Exclusion criteria the same as for study group

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will consist of 51 patients with masticatory muscle pain for at least 3 months, diagnosed on basis of DC/TMD protocol
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Relationship between masticatory muscle pain and polimorphism of serotonin receptor gene HTR2A - rs4941573 and dopamine receptor gene DRD3 - rs6280 | January 3, 2023 - January 3, 2024
  Each participant will undergo genetical blood test.
Relationship between masticatory muscle pain and serotonin and dopamine levels. | January 3, 2023 - January 3, 2024
  Each participant will undergo blood test.
Relationship between masticatory muscle pain and Gamma-aminobutyric acid (GABA), Tumor Necrosis Factor α (TNF-α), CGRP, SERT, interleukin 1B, interleukin 6, interleukin 8, interleukin 10 and interleukin 17A. | January 3, 2023 - January 3, 2024
  Each participant will undergo blood test.

SECONDARY OUTCOMES:
Relationship between masticatory muscle pain and depression assessed by Patient Health Questionnaire. | January 3, 2023 - January 3, 2024
  Each participant will fill in Patient Health Questionnaire - 9. PHQ-9 total score for the nine items ranges from 0 to 27.Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Relationship between masticatory muscle pain and PPTs. | January 3, 2023 - January 3, 2024
  Participants from study group will be tested using algometer to determine pressure pain threshold in masseter muscle and temporal muscle.
Relationship between masticatory muscle pain and anxiety assessed by Generalized Anxiety Disorder -7. | January 3, 2023 - January 3, 2024
  Each participant will fill in Generalized Anxiety Disorder -7 that consists of 7 items. Total score ranges 0-21 points. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Relationship between masticatory muscle pain and perceived stress assessed by Perceived Stress Scale. | January 3, 2023 - January 3, 2024
  Each participant will fill in Perceived Stress Scale -10. Scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items. It can range from 0 to 40. Scores ranging from 0-13 would be considered low stress,14-26 would be considered moderate stress, 27-40 would be considered high perceived stress.
Relationship between masticatory muscle pain and satisfaction with life assessed by Satisfaction With Life Scale. | January 3, 2023 - January 3, 2024
  Each participant will fill in Satisfaction With Life Scale which consist of five questions with 5 possible answers. Total score range is 35. Higher score represents higher life satisfaction. Score ranging from 5-9 as considered as extremly dissatisfied with life, 10-14 dissatisfied, 15-19 slightly dissatisfied, 20-24 slightly satisfied, 25-29 satisfied, 30-35 extremely satisfied.
Relationship between masticatory muscle pain and Type D personality assessed by DS-14 quesstionaire. | January 3, 2023 - January 3, 2024
  Each participant will fill DS-14 questionnaire which contains 14 Likert-style questions. Each questions has a score range of 0-4. This questionnaire consist of two subscales: negative affectivity and Social Inibition. A cut-off of 10 on both scales is used to classify subject as type-D personality. Maximum score in both scales is 28.
Relationship between masticatory muscle pain and coping with stress assessed by mini COPE. | January 3, 2023 - January 3, 2024
  Each participant will fill in mini COPE. Questionnaire consists of 28 statements that make up 14 stress coping strategies.Some testing strategies were divided into four categories and corresponding strategies (inventory scales): active coping (including: active coping, planning, positive reevaluation), helplessness (including: taking psychoactive substances, cessation of actions, blaming self), seeking support (including: seeking emotional support, seeking instrumental support), avoidance behaviors (including dealing with something else, denying, discharging). three strategies create independent factors (turning to religion, acceptance, sense of humor). The range of results for each statement ranges from 0 to 3 points. The calculation of the results consists in adding to each other points for the answers regarding two theorems that make up the given scale, and then dividing by 2.
Relationship between masticatory muscle pain and central sensitization assessed by Central Sensitization Inventory. | January 3, 2023 - January 3, 2024
  Each participant will fill in Central Sensitizatin Inventory. This questionnaire consist of two parts. First part includes 25 questions regarding common central sensitivity symptoms. It allows to categorize participant into one of five categories: subclinical (0-29), mild (30-39), moderate (40-49), severe (50-59), and extreme (60-100) Second part is not scored, but it determines if the participant has been diagnosed with certain CSS disorders or related disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland